CLINICAL TRIAL: NCT00675168
Title: PET/CT and Roentgen in Lung Cancer. Evaluation of Patients in General Practice
Brief Title: Positron Emission Tomography (PET)/Computed Tomography (CT) and Roentgen in Lung Cancer: Evaluation of Patients in General Practice
Acronym: PROLOG
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Mie Jung Nielsen, MD, Odense University Hospital, Department of Nuclear Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: PROLOG
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; PET/CT; Diagnosis
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: PET/CT (low-dose) — 400 mBq 18F-flour-deoxyglucose given iv. 60 min. before PET/CT-scan
  Other Names: FDG

SUMMARY:
The prognosis of lung cancer depends much on the stage of the disease at the time of diagnosis. Only 16 % of lung cancer can be offered curative intended surgery. Chest x-ray is the gate-keeper in lung cancer diagnosis, but it has a miss rate of 20-60 %. A false negative chest x-ray often causes prolonged delay in diagnosis - often months.

Recently a "48 hour diagnosis guaranty" has been implemented, which helps accelerate the system delay (delay from referral to diagnosis). But chest x-ray is still the gate-keeper; if the chest x-ray is negative further examination ceases.

PET/CT has a higher sensitivity (96 %), than chest x-ray. In the latter years only little improvement in the survival rate of lung cancer has been made. Screening studies is currently been performed, but it's time for innovative thinking. PET/CT has established its place in the staging of lung cancer. But studies like this may help to place PET/CT in the chain of examination making it more cost-beneficial.

The overall aim of this study is to improve patient course with earlier diagnosis of lung cancer.

DETAILED DESCRIPTION:
Background

Each year 3500 new patients in Denmark are diagnosed with lung cancer. This makes lung cancer the second most common cancer in Denmark. In Europe lung cancer is the most common cancer with an estimated 377 000 new cases each year. Lung cancer has a poor prognosis with a 5 year relative survival rate of approximately 10 % in Europe and 15 % in USA. The survival rate in Denmark has been inferior to that of other Nordic countries, partly because of unfavorable stage distribution at the time of diagnosis. Lately there has been an improvement in one year relative survival rate, because more patients are offered life prolonging chemotherapy, but with no influence on the 5-year survival rate.

The main investigation for suspected lung cancer is a chest x-rays, but chest x-rays has a miss rate of 20-60 %, which tends to delay the diagnosis by several months. Nodules < 1-1.6mm and centrally placed tumor increase the likelihood of a missed diagnosis.

Studies on screening for lung cancer has been promising, but has not yet shown an effect in terms of reduced mortality.

FDG-PET/CT is rapidly gaining acceptance in clinical oncology for diagnosing tumors, staging disease, and evaluating treatment response. PET/CT is a new scanner modality combinng the diagnostic accuracy of computed tomography (CT) with the metabolic activity recording of positron emission tomography (PET). A metaanalysis of PET alone has shown a sensitivity and specificity of 96 % and 78%, respectively with respect to diagnosis of pulmonary nodules. Studies with the combined PET/CT technique are expected to increase the specificity without affecting the high sensitivity.

False positive PET/CT scans are often due to increased uptake of 18F-flourdeoxyglucose (FDG) in inflammatory cells (granulomas, tuberculosis, chronic infection). False-negative PET/CT scans is often due to small size (< 5-7 mm) or high-differentiated malignancies (bronchio-alveolar carcinomas, carcinoids).

To our knowledge no similar study has been published or is currently under investigation.

Methods

The study is divided into 2 retrospective investigations (Pre-PROLOG 1 and 2) and a prospective study PROLOG.

Pre-PROLOG 1 We wish to identify high pretest likelihood of lung cancer based on the information from the referral to chest x-ray. All patients referred to a chest x-ray examination from General Practice between January 1 and March31, 2005, to the Department of Radiology, Odense University Hospital (OUH), in total 1201 patients. Referral diagnosis and information were registered in this retrospective survey.

Patients were two years later compared with patients in the Danish Lung Cancer Register (DLCR). DLCR is a national register, whereto 55 departments in Denmark report new cases of lung cancer. There is a certain overlap between reports, and an estimated 90 % of all lung cancer in Denmark are assumed registered in DLCR.

The data has been collected and is currently being analyzed. Preliminary results show that:

37 of our 1201 patients were registered in the Danish Lung Cancer Register on the October 17, 2007. Nine of the patients had been diagnosed prior to the chest x-ray and one patient was diagnosed as having a mesothelioma. Out of the 1192 referred to a chest x-ray under different diagnoses (without the 9 known lung cancers) 27 (2.2 %) turned out within the next 2 years to have lung cancer.

Pre-PROLOG 2 We wish to explore the delay in the diagnosis and treatment of lung cancer. All lung cancer patients diagnosed at Odense University Hospital (all Departments) between 1 January 2006 and 30 June 2007 are identified. A questionnaire is sent to all patients still alive, in which the patients among other things are asked about the time of their first symptom, 1st visit to their GP due to symptoms retrospectively related to lung cancer. Another questionnaire is sent to the patients' GP and finally, case records are examined. The delay is divided into patient delay (from first symptom to 1st visit to GP), doctor delay (from 1. visit to GP to referral to chest x-ray/hospital department) and system delay (from referral to start of treatment).

Questionnaires are expected to be sent out in December 2007.

PROLOG All patients complying with the inclusion criteria (age >50 years and suspicion of lung cancer, based on clinical symptoms and /or history with including being a current or former smoker and other risk factors laid down by the Pre-PROLOG 1 study) are referred to an ordinary chest x-ray at the Department of Radiology OUH. The same day or the next day a PET/CT scan is performed at the Department of Nuclear Medicine, OUH. All patients will have both a chest x-ray and a PET/CT-scan.

Following outcomes are possible following blind readings of both the chest x-ray and the PET/CT scan:

1. Patients with a suspicious chest x-ray: All have a chest CT scan and are referred to further examination at the Department of Medicine - Section of Lung Disease, OUH.
2. Patients with an unsuspicious chest x-ray: All go back to their GP to follow-up.
3. Patients with a positive PET/CT scan (intrathoracal): All are referred to further examination at the Department of Medicine - Section of Lung Disease.
4. Patients with a negative PET/CT scan: All are sent back to their GP for follow-up.
5. Patients with a negative intrathoracal PET/CT, but a positive extrathoracal PET/CT: Report with suggestion of further action is sent to the GP. Who refers the patient to further examination.

In all cases our Gold Standard is a malignant pathology diagnosis. The status of all patients is determined on entrance and at time 6 months, 12 months, and 24 months. Patients who do not have a positive pathology diagnosis after 24 month are regarded as not having lung cancer. The start of the main study is expected to start in the spring 2008.

Ethics

The study follows Helsinki Declaration II nr. 503 of 24 June 1992 and nr. 499 of 12 June 1996.

Possible positive effects by participating in the study:

* Early diagnosis of lung cancer, with a better chance of curative treatment/better prognosis
* Early diagnosis of other malignancies

Possible negative effects by participating in the study:

* A PET/CT gives an effective radiation dose of 14 mSv, which is comparable to approximately 4-5 times the background radiation in Denmark (3 mSV).
* Focus on illness and the possible following psykosociale effects

The positive advantages by participating in the study are thought to outweigh the negative consequences. It's up to the patient to access the possible effects of the study after thorough information fore and against. All participation is voluntarily. If patients do not want to participate, normal examination is carried out.

All informations are kept in agreement with the departmental order nr. 528 of 15 June 2000 chapter 1, 2 og 3 §§ 41-42.

ELIGIBILITY:
Inclusion Criteria:

* Pt. referred from general practice to a chest x-ray
* age 60-80 years
* current or former smoker

Exclusion Criteria:

* previously diagnosed with lung cancer
* contraindications to PET/CT

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1700 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of chest x-ray and PET/CT in Lung Cancer | min. two years of follow up

SECONDARY OUTCOMES:
Positive/negative predictive values of chest x-ray and PET/CT Operability - surrogate for survival Numbers of false positive PET/CT Numbers of false negative PET/CT Numbers of invasive procedures Cost-effectiveness | min. two years of follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of Nuclear Medicine, Odense, Funen
  - Odense, Fünen